CLINICAL TRIAL: NCT06641323
Title: Ozonized Gel vs Gaseous Ozone Against S. Mutans in Deciduos Molars Caries: Randomized Clinical Trial
Brief Title: Ozonized Gel vs Gaseous Ozone Against S. Mutans in Deciduos Molars Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-OZONECARIES
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone gel group (Experimental)
  Interventions: Other: Ozonized gel
- Gaseous ozone group (Active Comparator)
  Interventions: Device: Ozonized water

INTERVENTIONS:
Other: Ozonized gel — Administration of Ozonized Gel GeliO3
  Arms: Ozone gel group
Device: Ozonized water — Admininstration of Gaseous ozone (Healozone X4)
  Arms: Gaseous ozone group

SUMMARY:
The aim of this study is to verify, through bacteriological analysis, the efficacy of reducing the bacterial load referred to the presence of Streptococcus Mutans in carious lesions of viable deciduous molars by application of gaseous ozone or ozonized gel.

Patients who meet the eligibility criteria and for whom the legal guardians have signed the informed consent, will undergo treatment of the carious lesion with gaseous ozone or ozonized gel. After selective removal of dentin, a bacterial sample will be taken from the carious surface with a sterile paper cone at time T0; then ozone will be applied for 30 seconds, the surface will be washed with sterile saline and dried with air, a second sample will be taken at time T2; finally, ozone will be applied for another 30 seconds, the surface will be washed with sterile saline and dried with air, a third sample will be taken at time T2.

Patients are then randomised into two groups:

Test group: gaseous ozone (Healozone X4) is applied to the carious lesion for 30 seconds and then for another 30 seconds.

Control group: ozone gel (GeliO3) will be applied to the carious lesion for 30 seconds and then for another 30 seconds.

Changes in the following indices will be assessed at the first visit and when the samples are taken at T0, T1, T2: compliance assessment (FLACC scale), sensitivity test (Schiff Air Index), assessment of lesion severity and extent (ICDAS), assessment of gingival inflammation (GI), assessment of plaque index (PI), assessment of severity of enamel erosion (Bewe index).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from carious lesion on viable deciduous molar
* patients' compliance

Exclusion Criteria:

* patients with early loss of deciduous molars for carious lesions or orthodontic reasons
* non-viable deciduous molars
* deciduous molars with traumatic lesions

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Change in S. mutans counts | Baseline (T0), after 30 seconds (T1) and after 60 seconds (T2)
  Evaluation of Colony forming units (CFU) of bacterials samples after treatment.

SECONDARY OUTCOMES:
Change in FLACC | Baseline (T0), and after 60 seconds (T2)
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain for children with a score of 0 to 2 for each evaluation.
Change in Schiff Air Index | Baseline (T0), and after 60 seconds (T2)
  Scoring criteria:
  0.= the subject does not respond to air stimulation;
  1. = the subject responds to stimulation with air but does not require interruption;
  2. = the subject responds to stimulation with air and requests interruption or moves away from the stimulus;
  3. = the subject responds to stimulation with air, considers the stimulus painful, requests its interruption or moves away from it.
Gingival Index (calculated on Ramfjiord teeth) | Baseline (T0)
  Scoring criteria:
  0 = normal gingiva, no inflammation, no erythema, no bleeding
  1. = mild inflammation, slight erythema, minimal superficial alterations, no bleeding
  2. = moderate inflammation, erythema, bleeding on probing
  3. = severe inflammation, severe erythema and swellling, tendency to spontaneous bleeding, possible ulcers
Plaque Index (calculated on Ramfjiord teeth) | Baseline (T0)
  Scoring criteria:
  0 = no plaque
  1. = thin layer of plaque at the gingival margin, detectable only by scraping with a probe
  2. = moderate layer of plaque along the gingival margin; free interdental spaces, but plaque is visible to the bare eye
  3. = abundant plaque along the gingival margin; plaque-filled interdental spaces.
ICDAS | Baseline (T0)
  Scoring criteria:
  0 = healthy
  1. = White/brown stain in dry enamel
  2. = White/brown stain on wet enamel
  3. = Microcavity in dry enamel <0.5 mm with no visible dentin
  4. = Dark dentin shade seen through wet enamel with or without microcavity
  5. = Dentin exposure in the cavity> 0.5 mm in the middle of the dry tooth surface
  6. = Dentin exposure in cavity greater than half of the tooth surface
Basic Erosive Wear Examination | Baseline (T0)
  Scoring criteria:
  0 = no tooth erosion
  1. = superficial enamel loss
  2. = hard tissue loss involving < 50% of tooth surface
  3. = hard tissue loss involving > 50% of tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.